CLINICAL TRIAL: NCT05052944
Title: Single-sided Deafness and Cochlear Implantation
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00230644
Record Dates: First submitted 2021-09-14; First posted 2021-09-22 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Unilateral; Hearing Loss, Sudden; Hearing Loss, Cochlear; Hearing Loss in Left Ear; Hearing Loss in Right Ear; Labyrinthitis
Keywords: cochlear implantation
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Sensorineural; Hearing Loss, Unilateral; Hearing Loss, Sudden; Labyrinthitis | interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cochlear implant recipients: Patients with single-sided deafness undergoing cochlear implantation
  Interventions: Device: Cochlear implantation

INTERVENTIONS:
Device: Cochlear implantation — Patients who receive cochlear implant for single-sided deafness
  Other Names: Med El cochlear implant

SUMMARY:
This observational study evaluates the effects of cochlear implantation in patients with deafness in one ear.

DETAILED DESCRIPTION:
Cochlear implant (CI) technology has been widely used for individuals with bilateral sensorineural hearing loss to improve the ability to perceive sound by bypassing the damaged portion of the inner ear. Recently in the U.S., Cochlear implantation has also been approved by the FDA for treatment of single-sided deafness. By restoring binaural hearing, cochlear implantation in unilateral hearing loss may improve hearing in noise and sound localization, however its audiologic outcomes and quality of life impact for patients remain incompletely understood.

This study aims to establish a prospective database to track and quantify the change in general health status, tinnitus severity, spatial hearing ability, and difficulty with communication in noise after unilateral cochlear implantation in patients with SSD undergoing routine medical and audiologic evaluation at the Johns Hopkins Cochlear Implant Center. Study participants will complete survey questionnaires and undergo standard-of-care audiological evaluation before and after cochlear implantation. Data collected in this study will be invaluable in gaining an in-depth understanding of the effects of cochlear implantation in patients with SSD in the context of current FDA guidelines, and lead to better counseling and patient selection for this treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* For individuals ages 18 years-old and above, limited benefit from unilateral amplification is defined by test scores of 5% correct or less on monosyllabic consonant-nucleus-consonant (CNC) words in quiet when tested in the ear to be implanted alone.
* Before implantation with a cochlear implant, individuals with SSD or AHL must have at least 1-month experience wearing a Contra Lateral Routing of Signal (CROS) hearing aid or other relevant device and not show any subjective benefit.
* Medical and surgical clearance for cochlear implantation.

Exclusion Criteria:

* Not meeting FDA candidacy criteria for cochlear implantation in SSD
* Inability to perform audiologic tasks (e.g. non-English speaking)
* Medical or surgical contraindication to general anesthesia or cochlear implant surgery
* Does not wish to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises individuals with single-sided deafness or asymmetric hearing loss resulting in poor hearing in one ear.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-11-09 (Actual)

PRIMARY OUTCOMES:
Change in Speech recognition in quiet | Baseline and up to 1 year post-implantation
  Change in Speech recognition in quiet will be assessed using the percent correct on Consonant-Noun-Consonant words and phonemes.
Change in Speech recognition in noise | Baseline and up to 1 year post-implantation
  Change in Speech recognition in noise will be assessed using the percent correct on AzBio with multitalker babble at 8dB signal-to-noise ratio.

SECONDARY OUTCOMES:
Change in Spatial hearing as assessed by the Spatial Hearing Questionnaire | Baseline and up to 1 year post-implantation
  Score on Spatial Hearing Questionnaire. Range: 0-100. Higher score signifies less handicap related to sound localization.
Change in Tinnitus handicap as assessed by the Tinnitus Handicap Inventory | Baseline and up to 1 year post-implantation
  Score on Tinnitus Handicap Inventory. Range: 0-100. Higher score signifies more handicap due to tinnitus.
Change in Hearing aid benefit as assessed by the Abbreviated Profile of Hearing Aid Benefit | Baseline and up to 1 year post-implantation
  Score on Abbreviated Profile of Hearing Aid Benefit. Range: 0-100. Higher score signifies more frequent problems with hearing.
Change in Health utility as assessed by the Health Utility Index | Baseline and up to 1 year post-implantation
  Score on Health Utility Index. Range: 0-1.0. Lower score signifies lower health utility.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Sun, MD, Principal Investigator — JHU
Locations (5):
- United States (5):
  - Johns Hopkins Bayview, Baltimore, Maryland
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Johns Hopkins Suburban, Bethesda, Maryland
  - Johns Hopkins Greenspring Station, Lutherville-Timonium, Maryland
  - Johns Hopkins White Marsh, Nottingham, Maryland

IPD SHARING:
Plan to Share IPD: No